CLINICAL TRIAL: NCT02126553
Title: Phase II Study of Lenalidomide Maintenance in Patients With High Risk AML in Remission
Brief Title: Lenalidomide in Treating Patients With High Risk Acute Myeloid Leukemia in Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0116; NCI-2014-01176 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0116 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Alkylating Agent-Related Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lenalidomide) (Experimental): Patients receive lenalidomide PO QD on days 1-28. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lenalidomide

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This phase II trial studies how well lenalidomide works in treating patients with acute myeloid leukemia that have had a decrease in or disappearance of signs and symptoms of cancer, although cancer still may be in the body and may be likely to come back or spread. Biological therapies, such as lenalidomide, use substances made from living organisms that may kill cancer cells by blocking blood flow to the cancer and by stimulating white blood cells to kill the cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess relapse-free survival (RFS) of patients with acute myeloid leukemia (AML) treated with lenalidomide maintenance therapy after achieving remission.

SECONDARY OBJECTIVES:

I. To assess overall survival (OS) of patients with AML treated with lenalidomide maintenance.

II. To assess event-free survival (EFS) of patients with AML treated with lenalidomide maintenance.

III. To assess the duration of remission (CRd) of patients with AML treated with lenalidomide maintenance.

IV. To assess toxicity and safety of lenalidomide maintenance in patients with AML.

V. To assess the effects of lenalidomide maintenance on natural killer (NK) cell modulation and dynamics of minimal residual disease and their relationship to outcomes.

OUTLINE:

Patients receive lenalidomide orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 55 years with high risk AML who have achieved their FIRST complete remission (CR) or complete remission with incomplete recovery (CRi) within 12 months of enrollment and are not immediately candidates for allogeneic stem cell transplant; patients above age 55 who are not eligible for other protocols may be considered for enrollment on a case by case basis after discussion with the principal investigator (PI)
* Patients in their FIRST CR or CRi may be eligible for enrollment only if they have a high risk feature, including, but not limited to: adverse karyotype, fms-related tyrosine kinase 3 (FLT3) mutation, history of antecedent hematologic disorder (AHD), presence of dysplasia in the bone marrow, therapy-related AML, history of requiring more than 1 cycle of intensive induction chemotherapy to achieve first remission, or presence of persistent minimal residual disease (detected by cytogenetics, molecular markers, or flow cytometry) at any point after initial induction cycle; patients aged >= 18 years with AML who have achieved a SECOND CR or CRi within 12 months of enrollment and are not immediately candidates for allogeneic stem cell transplant are also eligible
* Patients should have received induction chemotherapy for AML and at least 1 consolidation
* Patients with history of extramedullary AML, except for central nervous system (CNS) involvement that is currently controlled, will not be eligible for enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status of < or = 3
* Serum total bilirubin < or = to 1.5 X the upper limit of normal (ULN)
* Serum creatinine < or = to 2.5 x ULN
* Absolute neutrophil count (ANC) > 0.5 x 10^9/L
* Platelet count > or = 30 x 10^9/L
* For females of childbearing age, they may participate it they: a. have a negative serum or urine pregnancy test within 10 to 14 days of enrolling (a second pregnancy test will be performed within 24 hours (hrs) of starting therapy and both negative pregnancy tests will be required for starting therapy); b. agree to either abstinence or 2 effective contraceptive methods throughout the treatment period and up to 28 days after discontinuing treatment
* For male patients with a female partner of childbearing age, they may participate if they agree to either abstinence or 2 effective contraceptive methods throughout the treatment period and up to 28 days after discontinuing treatment
* All study participants be willing and able to comply with the requirements of the Risk Evaluation and Mitigation Strategies (REMS) program
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS program
* Ability to understand and sign informed consent

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (APL), AML - M3 by French American British (FAB) classification based on morphology, immunophenotype, molecular, or cytogenetics studies
* Diagnosis of AML associated with the following karyotypes: inversion (inv)(16), t(16;16), t(8;21), t(15;17), or t(9;22)
* Uncontrolled intercurrent illness including, but not limited to ongoing or active uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Previous treatment with lenalidomide for AML
* Patients with documented hypersensitivity to any components of the study program
* Females who are pregnant
* Patients with active CNS disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-11-13 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tapan M Kadia, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: November 2014 to November 2021
Period: Overall Study
Arm/Group | Treatment (Lenalidomide)
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Lenalidomide)
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 59 [23 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 20
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Relapse-free Survival (RFS)
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 7 Years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Lenalidomide)
Number analyzed (Participants) | 29
Months | 21.5 [0.7 to 54.3]

2. Secondary Outcome: Overall Survival (OS)
Description: Time from date of treatment start until date of death due to any cause or last Follow-up. Survival will be measured by the estimated median survival computed by Kaplan-Meier (K-M) analysis, which is the time point at which the cumulative survival drops below 50%, if present. If not present then the median Overall Survival is not reached and not available (NA) as there are an insufficient number of participants with events. In either case ranges are provided for observed survival intervals used in the K-M analysis.
Time Frame: Up to 7 Years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Lenalidomide)
Number analyzed (Participants) | 29
Months | NA [1.3 to 54] — Median not reached due to insufficient number of participants with events.

3. Secondary Outcome: Event-free Survival (EFS)
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse, death or discontinuation due to adverse events.
Time Frame: Up to 7 Years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Lenalidomide)
Number analyzed (Participants) | 29
Months | 12 [0.5 to 54.3]

4. Secondary Outcome: Complete Response (CR) Duration
Description: Complete Response is defined as disappearance of all clinical and/or radiologic evidence of disease, including extramedullary leukemia. Neutrophil count >/= 1.0 x 10^9/L and platelet count>/= 100 x 10^9, and bone marrow differential showing </=5%blasts. Response date to loss of response or last follow up. Remission duration will be measured by the estimated median remission duration computed by Kaplan-Meier (K-M) analysis, which is the time point at which the cumulative remission duration drops below 50%, if present. If not present then median remission duration is not reached and not available (NA) as there are an insufficient number of participants with events. In either case ranges are provided for observed survival intervals used in the K-M analysis.
Time Frame: Up to 7 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Lenalidomide)
Number analyzed (Participants) | 29
Months | NA [0.7 to 54.3] — Median not reached due to insufficient number of partcipants.

ADVERSE EVENTS:
Time Frame: Up to 7 years
Arm/Group | Treatment (Lenalidomide)
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 7/29
Other Adverse Events (participants affected / at risk) | 22/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide) (N=29)
Cellulitis Hand (Infections and infestations) | 1 (1)
elevated transaminases (Metabolism and nutrition disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Cellulitis Foot (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide) (N=29)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (2)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
Itchy Scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 2 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6 (6)
Heartburn/dyspepsia (Gastrointestinal disorders) | 4 (4)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10^ (Infections and infestations) | 1 (1)
Foot Cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia Back and Neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (inflammation/damage of muscle) (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Neuropathy: motor (Nervous system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 4 (4)
Headache (General disorders) | 2 (2)
back pain (General disorders) | 1 (1)
Platelets Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 12 (12)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Vision-photophobia (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT02126553/Prot_SAP_000.pdf